CLINICAL TRIAL: NCT00344409
Title: A Double-blind, Placebo Controlled, Randomized Study of KRN321 for the Treatment of Anemia in Cancer Patients
Brief Title: A Double-blind Study of KRN321 for the Treatment of Anemia in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KRN321-SC/05-A54
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Anemia
Keywords: darbepoetin alfa; anemia; cancer patients; platinum containing chemotherapy
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa

SUMMARY:
To compare the effectiveness of KRN321 to placebo in the treatment of anemia in cancer patients receiving multi cycle platinum-containing chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as lung or gynecological cancer
* patients receiving platinum containing chemotherapy
* written informed consent
* hemoglobin concentration less than 11 d/dL at enrollment
* life expectancy of more than 4 months

Exclusion Criteria:

* hemolysis, gastrointestinal bleeding, postoperative bleeding
* iron deficiency
* megaloblastic anemia
* any primary hematological disorder that could cause anemia
* received > 2 RBC transfusions with 4 weeks or any RBC transfusion within 2 weeks before randomization
* prior treatment with KRN321
* received erythropoetin therapy within 8 weeks before treatment

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-03; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To compare the proportion of subjects who reach red blood cell transfusion trigger

SECONDARY OUTCOMES:
To compare the effectiveness of KRN321 on the proportion of subjects achieving hemoglobin response
To compare the proportion of subjects who receive red blood cell transfusions
To compare the effectiveness of KRN321 based on quality of life scores

CONTACTS AND LOCATIONS:
Overall Officials: Nagahiro Saijo, MD, Study Chair — National Cancer Center Hospital East
Locations (7):
- Japan (7):
  - Shikoku region, Ehime
  - Kyusyu region, Fukuoka, Kagoshima
  - Chugoku region, Hiroshima, Tottori
  - Tohoku region, Iwate, Miyagi
  - Kinki region, Nara, Osaka, Hyogo
  - Tokai region, Shizuoka, Aichi
  - Kanto region, Tokyo, Chiba, Ibaraki, Saitama, Niigata